CLINICAL TRIAL: NCT02072629
Title: Healthy Child Uganda: Can Village Health Volunteers Trained in Integrated Community Case Management of Childhood Illness Improve Access to Care for Africa's Most Vulnerable Children?
Brief Title: HCU: Can VHVs Trained in ICCM Improve Care for Children
Acronym: HCU:VHV/ICCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jennifer L. Brenner, Clinical Associate Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: E-22746
Record Dates: First submitted 2014-02-21; First posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Diarrhoea; Pneumonia; Malaria
Keywords: Antimalarials; Antibiotics; ORS Zn; Village Health Volunteers; Integrated Community Case Management
MeSH Terms: conditions — Diarrhea; Pneumonia; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Training of VHVs in iCCM (Experimental): In these villages VHVs will be provided with iCCM training and equipped to support iCCM in their villages
  Interventions: Other: Training of VHVs in iCCM

INTERVENTIONS:
Other: Training of VHVs in iCCM — Village Health Volunteers will be trained in Integrated Community Case Management (iCCM) of childhood illness

SUMMARY:
This study will assess how the current VHV (VHV=CHW, community health worker) scope can be expanded to include iCCM and if such group interventions can provide improved access to treatment for children.

In rural SW Uganda, can iCCM provided by lay volunteers, increase the proportion of children with diarrhoea receiving ORS/Zn, ARI receiving anti-biotics, and fever/malaria receiving anti-malarials?

ELIGIBILITY:
Inclusion Criteria:

* Women living in intervention and comparison villages
* Mother to at least one child under 59 months old

Exclusion Criteria:

-No living child

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4071 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Absolute change pre/post intervention (VHV ICCM training) in proportion of U5s receiving (a) antimalarial for fever (b) ORS/Zn for diarrhea (c) Abx for pneumonia | pre- (Dec 2010) post- (Dec 2012) intervention (2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Maling, MD, Principal Investigator — Mbarara University of Science and Technology; jenn Brenner, MD, Study Director — University of Calgary

REFERENCES:
- [Derived] Oliphant NP, Manda S, Daniels K, Odendaal WA, Besada D, Kinney M, White Johansson E, Doherty T. Integrated community case management of childhood illness in low- and middle-income countries. Cochrane Database Syst Rev. 2021 Feb 10;2(2):CD012882. doi: 10.1002/14651858.CD012882.pub2. PMID 33565123